CLINICAL TRIAL: NCT06480461
Title: A Phase Ⅰb/Ⅱ Study to Evaluate the Tolerability, Safety, and Efficacy of VGN-R09b in Patients With Parkinson's Disease
Brief Title: A Trial to Evaluate Safety and Efficacy of a Product Named VGN-R09b in Patients With Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGN-R09b-101
Record Dates: First submitted 2024-06-14; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Parkinson's Disease
Keywords: VGN-R09b
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8.0×10^11 vg (Experimental): 3 subjects on 8.0×10^11 vg for at least 4 weeks post infusion
  Interventions: Drug: VGN-R09b
- 1.6×10^12 vg (Experimental): 3 subjects on 1.6×1012 vg for at least 4 weeks post infusion
  Interventions: Drug: VGN-R09b
- 3.2×10^12 vg (Experimental): 3 subjects on 3.2×1012 vg for at least 4 weeks post infusion
  Interventions: Drug: VGN-R09b

INTERVENTIONS:
Drug: VGN-R09b — This is a Phase I/II trial, with safety as the primary measure. Sample size is not determined through statistical justification. There will be 3 subjects in each dose cohort in the dose escalation part. In the dose expansion part, a sham surgery group and 2 dose groups will be designed; 10 subjects will be enrolled in each group.

SUMMARY:
A phase Ⅰ/Ⅱ study to evaluate the tolerability, safety, and efficacy of VGN-R09b in pa-tients with Parkinson's disease

DETAILED DESCRIPTION:
In the open-label dose escalation part, 3 dose cohorts will be explored, with 3 subjects per cohort.

Cohort 1: 3 subjects on 8.0×10^11 vg for at least 4 weeks post infusion Cohort 2: 3 subjects on 1.6×10^12 vg for at least 4 weeks post infusion Cohort 3: 3 subjects on 3.2×10^12 vg for at least 4 weeks post infusion In the dose-escalation part, each cohort follows the principle of sentinel administration (i.e., one subject will be enrolled and dosed first in each cohort). If no significant safety risk is observed within 4 weeks after administra-tion, the remaining 2 subjects will be dosed.

Additional cohort(s) and/or a safe low and high dose will be determined by the safety review committee (SRC) to initiate Part II

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria:

  1. Male or female, ≥40 years and <75 years of age at Screening.
  2. Diagnosis of Idiopathic Parkinson's disease according to the UK Brain Bank.
  3. Insufficient control of motor symptoms with an average of ≥2.5 hours of OFF time per day over 3 consecu-tive days despite optimized treatment, as confirmed by the PD patient diary at Screening.
  4. Stable Parkinson's symptoms and an optimal regimen of Parkinson's medications for at least 4 weeks prior to screening, with a duration of levodopa treatment of ≥1 year.
  5. Hoehn and Yahr Stage 2.5~4 on "off" state.
  6. All men and women of childbearing potential must be willing to use at least one highly effective method of contraception from the signing of informed consent until one year after administration of the study drug.
  7. Men must agree not to donate sperm, and women must agree not to donate eggs within at least one year after administration of the study drug.
  8. The patient must understand the purpose and risks of the study, sign and date the informed consent, and give authorization to use the protected health information in accordance with national and local privacy regulations.
  9. The patient has a reliable study partner/informant (e.g., a family member, friend) willing and able to partici-pate in the study as a source of information on the patient's health status and cognitive and functional abili-ties (including providing input into the rating scales).

Exclusion Criteria:

* Subject has any of the following diseases or disease history

  1. Atypical or secondary parkinsonism, including but not limited to symptoms believed to be due to trauma, brain tumor, infection, cerebrovascular disease, or other neurological disease, or to drugs, chemicals, or tox-ins, as determined by the Investigator.
  2. Known pathogenic gene mutations of GBA1, PINK1, and Parkin
  3. MoCA score ≤16
  4. Currently active infection or a severe infection (e.g., pneumonia, septicemia, central nervous system infec-tions [e.g. meningitis, encephalitis]) within 12 weeks prior to Screening
  5. Active infection of HBV, HCV or TP, or with HIV-positive at screening.
  6. Unstable autoimmune disease within 6 months prior to Screening, or requiring chronic immunosuppression.
  7. Poorly controlled diabetes (Screening glycosylated hemoglobin [HbA1C] ≥ 7%), or uncontrolled hyperten-sion.
  8. History of stroke or transient ischemic attack, unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV), or clinically significant conduction abnormalities (e.g., un-stable atrial fibrillation) within 1 year prior to Screening.
  9. New or unstable psychiatric conditions (e.g. psychosis, severe depression, or with current suicidal ideation or suicide attempt) within 1 year of screening.
  10. History of malignancy within 3 years of screening, other than fully excised non-melanoma skin cancers, non-metastatic prostate cancer, and fully treated carcinoma in situ, provided it has been stable for at least 6 months.
  11. Any medical conditions that, in the opinion of the Investigator, could interfere with study-related proce-dures (including the safe performance of intraparenchymal injection), such as severe dyskinesia/impulse control disorders/tremor that may interfere with drug injection, brain implants, bleeding diathesis, clinically significant coagulopathy, thrombocytopenia, or increased intracranial pressure.

      Subject who is receiving or has a history of any of the following medications
  12. Any type of prior gene or cell therapy.
  13. Prior brain surgery for deep brain stimulation, focused ultrasound, infusion therapies or any other brain sur-gery for PD, or planned brain surgery for PD within 1 year after study entering.
  14. Any anticoagulant or antiplatelet therapies that could not be stopped before study drug injection.
  15. Any live vaccine within 4 weeks prior to Screening. Subject who meets any of the following test endpoints at screening
  16. An MRI showed a significant structural abnormality or lesion, bleeding, or >1 cm3 infarct, which, in the opinion of the Investigator, are contraindications to intraparenchymal injection.
  17. Clinically significant abnormalities in laboratory test values at Screening are in the opinion of the Investiga-tor, unsuitable for enrollment immediately.

      Subject under any of the following general conditions
  18. Contraindications to MRI/PET and/or agents used in PET.
  19. Contraindications to general anesthesia or deep sedation.
  20. Woman who is pregnant or breastfeeding.
  21. Participation within 3 months prior to Screening in another therapeutic investigational drug or device study, unless it can be documented that the patient received a placebo.
  22. Presence of substance (drug, alcohol) abuse within 2 years prior to Screening.
  23. The patient is generally frail or has any condition for which, in view of the Investigator, participation in the study would not be in the best interest of the patient or is likely to prohibit further participation during the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs)Vital signs | up to Week 52
  Vital signs, physical examination, laboratory test will be monitored after drug injection

SECONDARY OUTCOMES:
Changes in clinical outcomes | up to Week 52
  Subject number of MDS-Unified Parkinson's Disease Rating Scale Part I, II, III, and IV (UPDRS III) scores in ON- and OFF state；
Changes in clinical outcomes | up to Week 52
  Subject number of Levodopa equivalent daily dose (LEDD)；
Immunogenicity after injection | up to 52 weeks
  Subject number with positive antibodies of AAV9/AADC/Glial Cell Line-Derived Neurotrophic Factor (GDNF) in blood would be reported

IPD SHARING:
Plan to Share IPD: No